CLINICAL TRIAL: NCT02533713
Title: Effects of Exoskeleton-Assisted Gait Training on Bone Health and Quality of Life: A Randomized Clinical Trial
Brief Title: Effects of Exoskeleton-Assisted Gait Training on Bone Health and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Craig Hospital (Other)
Collaborators: Worcester Polytechnic Institute (Other); Massachusetts General Hospital (Other); University of Colorado, Denver (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Leslie Morse, Medical Director of Research, Craig Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001535
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Osteoporosis
Keywords: rehabilitation; bone strength; quality of life
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Immediate gait training (Experimental): Participants assigned to this arm will begin Exoskeleton assisted gait training right away and will continue training for the first 6 months of the study.
  Interventions: Device: Exoskeleton assisted gait training
- Delayed gait training (Other): Participants assigned to this arm will not gait train for 6 months. They will engage in Exoskeleton assisted gait training for the last 6 months of the study.
  Interventions: Device: Exoskeleton assisted gait training

INTERVENTIONS:
Device: Exoskeleton assisted gait training — Gait training will be performed 3 times a week for about an hour for 26 weeks. Gait training will be performed by a trained clinical physical therapist. The goal is to achieve 1 hour of continuous walking on a flat surface per training session. Gait training will continue for 26 weeks (78 sessions).

SUMMARY:
This is a randomized clinical trial to quantify the effects of exoskeleton-assisted gait on the musculoskeletal system and health-related quality of life.

DETAILED DESCRIPTION:
Investigators will test if exoskeleton-assisted ambulation confers skeletal benefits in a dose-dependent fashion. Investigators also will test if reintroduction of ambulation will be associated with improvements in quality of life due to improvements in mood, pain, and functional connectivity of emotional networks in the brain.

ELIGIBILITY:
Inclusion Criteria:

* 3 years or more after injury,
* Non-ambulatory AIS A-D spinal cord injury (C7-T12),
* 158-188 centimeters tall,
* Weigh less than 100 kilograms,
* Have a Modified Ashworth Scale (MAS) score of less than 3 in both lower extremities, and
* Have sufficient upper body strength to complete sit to sit transfers.
* Women of childbearing potential must agree to use contraceptive measures during participation in the study. They also will be required to have a negative pregnancy test (urine or serum) before receiving an imaging studies.

Exclusion Criteria:

* Current enrollment in another clinical trial
* Pregnancy
* Anyone with an initial blood pressure>140/90 mmHg, orthostatic hypotension with symptomatic fall in blood pressure >30 mmHg when upright,
* An active grade 2 or greater pressure ulcer that can be worsened by walking in the device,
* Lower extremity contractures that interfere with the ability to wear the device,
* An unhealed limb or pelvic bone fracture history of other neurological disease (e.g. stroke, peripheral neuropathy, myopathy),
* Active treatment for epilepsy,
* Current use of medications potentially affecting bone health (bisphosphonates, androgenic steroids, estrogenic steroids, lithium, glucocorticoid use for more than 3 months).
* Subjects with MRI-incompatible implants, pumps, or neurostimulators will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in tibial stiffness | baseline, six months, and 12 months
  assessed by finite element analysis of quantitative cat scan (QCT) of the knee

SECONDARY OUTCOMES:
Change in bone Volume | baseline, six months, and 12 months
  quantitative cat scan of the knee
Change in mood | baseline, six months, and 12 months
  Patient Health Questionnaire-9
Change in pain | baseline, six months, and 12 months
  International Spinal Cord Injury Basic Pain Data Set
Change in cortical activity | baseline, six months, and 12 months
  assessed by brain magnetic resonance imaging (MRI)
Change in health-related quality of life | baseline, six months, and 12 months
  psychological domain of the World Health Organization Quality-of-Life Scale (WHOQOL-BREF)

OTHER OUTCOMES:
Change in bone formation | baseline, six months, and 12 months
  assessed by circulating osteocalcin level
Change in marrow adiposity | baseline, six months, and 12 months
  Assessed by quantitative cat scan of the knee
change in bone resorption | baseline, six months, and 12 months
  assessed by circulating c-telopeptide level

CONTACTS AND LOCATIONS:
Overall Officials: Leslie R Morse, DO, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kowalski JL, Nguyen N, Battaglino RA, Falci SP, Charlifue S, Morse LR. miR-338-5p Levels and Cigarette Smoking are Associated With Neuropathic Pain Severity in Individuals With Spinal Cord Injury: Preliminary Findings From a Genome-Wide microRNA Expression Profiling Screen. Arch Phys Med Rehabil. 2022 Apr;103(4):738-746. doi: 10.1016/j.apmr.2021.09.005. Epub 2021 Oct 27. PMID 34717922